CLINICAL TRIAL: NCT04838704
Title: Ruxolitinib With Calcineurin Inhibitor and Methotrexate vs. Calcineurin Inhibitor Plus Methotrexate and Mycophenolate Mofetil as Graft Versus Host Disease Prophylaxis for HLA-haploidentical Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); Yinzhou Hospital Affiliated to Medical School of Ningbo University (Other); Ruijin Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCMvsCM
Record Dates: First submitted 2021-04-05; First posted 2021-04-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Graft Versus Host Disease
Keywords: Graft Versus Host Disease; ruxolitinib; HLA-haploidentical hematopoietic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RUX group (Experimental)
  Interventions: Drug: Ruxolitinib+Calcineurin inhibitor+Methotrexate
- Control group (Active Comparator)
  Interventions: Drug: Calcineurin Inhibitor+Methotrexate+Mycophenolate mofetil

INTERVENTIONS:
Drug: Ruxolitinib+Calcineurin inhibitor+Methotrexate — low-dose ruxolitinib combine with calcineurin inhibitor and short course of methotrexate.
  Arms: RUX group
Drug: Calcineurin Inhibitor+Methotrexate+Mycophenolate mofetil — calcineurin inhibitor and short course of methotrexate and mycophenolate mofetil
  Arms: Control group

SUMMARY:
Low Dose Ruxolitinib with Calcineurin Inhibitor and Methotrexate vs. Calcineurin Inhibitor plus Methotrexate and Mycophenolate mofetil as Graft Versus Host Disease prophylaxis for HLA-haploidentical hematopoietic stem cell transplantation in low-dose antithymocyte globulin (ATG) system.

DETAILED DESCRIPTION:
The is a prospective, randomized two-arm, and multicenter study. To compare the efficacy and safety of low-dose ruxolitinib combined with calcineurin inhibitor and methotrexate vs. calcineurin inhibitor plus methotrexate and mycophenolate mofetil as graft versus host disease prophylaxis for HLA-haploidentical hematopoietic stem cell transplantation in low-dose antithymocyte globulin (ATG) system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be diagnosed with malignant hematological disease.
2. aged 12-70 years.
3. Received HLA-haploidentical hematopoietic stem cell transplantation.
4. received myeloablative conditioning
5. Karnofsky score ≥70.
6. creatinine clearance ≥60 mL/min (according to the Cockcroft-Gault formula). (7) liver and kidney function: aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of the normal range (ULN), total bilirubin ≤ 2 × ULN; serum creatinine ≤ 1.5 × ULN.

8) left ventricular ejection fraction (LVEF) ≥ 50% on echocardiography (ECHO). 9) life expectancy >12 weeks. 10) Voluntarily signed the consent form and could understand and comply with the requirements of the study.

Exclusion Criteria:

1. Active autoimmune disease, such as SLE, rheumatoid arthritis, etc.
2. Current clinically significant active cardiovascular disease such as uncontrolled arrhythmia, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by New York Heart Association (NYHA) functional class, or a history of myocardial infarction within 6 months prior to enrollment.
3. Other serious medical conditions that may limit the patient's participation in this trial (e.g., progressive infection, uncontrolled diabetes).
4. human immunodeficiency virus (HIV) infection.
5. cirrhosis of the liver, active hepatitis.
6. Pregnant or lactating women.
7. Patients who are concurrently enrolled in any clinical trials of similar drugs.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
100-day cumulative II-IV aGVHD incidence after HSCT | From the date of transplantation to the first occurrence of grade II-IV acute GVHD, assessed up to 100 days.
  Cumulative incidence of grade II-IV acute GVHD occurring within the first 100 days following transplantation.

SECONDARY OUTCOMES:
Cumulative Incidence of Chronic GVHD | From the date of transplantation to the first diagnosis of chronic GVHD, assessed up to 3 years.
  The cumulative incidence of chronic GVHD following transplantation.n
Overall Survival | From the date of transplantation until death from any cause, assessed up to 3 years.
  Overall survival following is defined as the time from transplantation to death from any cause.
Adverse Events | From the date of transplantation to day 180 post-transplantation.
  Incidence and type adverse events following transplantation.
Cumulative Incidence of Relapse | From the date of transplantation to the first documented relapse, assessed up to 3 years.
  Cumulative incidence of disease relapse following transplantation is defined as the time from transplantation to the first documented disease recurrence.
GVHD-Free, Relapse-Free Survival | From the date of transplantation to the first occurrence of grade III-IV acute GVHD, systemic therapy-requiring chronic GVHD, relapse, or death, assessed up to 3 years.
  GVHD-free, relapse-free survival is defined as the time from transplantation to the first occurrence of grade III-IV acute GVHD, chronic GVHD requiring systemic therapy, disease relapse, or death from any cause.
Non-Relapse Mortality | From the date of transplantation to death without prior relapse or disease progression, assessed up to 3 years.
  Non-relapse mortality is defined as death without evidence of relapse or progression of the primary disease following transplantation.
Relapse-Free Survival | From the date of transplantation to the first documented relapse or death from any cause, assessed up to 3 years.
  Relapse-free survival is defined as the time from transplantation to the first documented relapse of the underlying disease or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No